CLINICAL TRIAL: NCT05821894
Title: Carotid Plaque Imaging Project (Identification of Vulnerable Atherosclerotic Plaques With Imaging and Biological Markers)
Brief Title: Carotid Plaque Imaging Project (CPIP)
Acronym: CPIP
Status: Recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Region Skåne (Unknown); The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other); Skåne University Hospital funds (incl. the Medical Training and Research Agreement/ALF) (Unknown); Swedish Foundation for Strategic Research (Other)
Responsible Party: Sponsor
Other Study IDs: CPIP
Record Dates: First submitted 2023-03-21; First posted 2023-04-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Atherosclerosis; Atherosclerotic Plaque
MeSH Terms: conditions — Atherosclerosis; Plaque, Atherosclerotic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, plaque, images
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Carotid Plaque Imaging Project (CPIP)
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study

SUMMARY:
The rupture or erosion of an atherosclerotic plaque with thrombosis or embolization often underlie heart attacks and strokes. The early identification of patients with atherosclerotic plaques prone to rupture or erosions, vulnerable plaques (VP), and their treatment before the occurrence of events is, therefore, one of the greatest cardiovascular challenges today. Possible approaches for early detection of VP include imaging techniques allowing visualization of plaque structure, circulating biomarkers and better understanding of the pathophysiologic mechanisms of the disease. In the carotid plaque imaging project the investigators study human atherosclerotic plaques (that are removed by endarterectomy) to disclose their underlying structure and mechanisms, finding possible novel therapeutic targets or markers for VP. The investigators also study plaque structure with imaging methods and try to develop new ways to detect VP using circulating or imaging markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old, male or female that are eligible for carotid endarterectomy due to atherosclerosis and that can provide informed consent.

Exclusion Criteria:

* Patients younger than 18 years old that cannot provide informed consent; pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with carotid stenosis undergoing endarterectomy at Skåne University Hospital (SUS), Malmö, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2005-10-26 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants suffering post-operative cardiovascular events (by 2025) | Follow up assessment year 2025 (recording of events occurring since 2023)
  Post-operative myocardial infarction, stroke, transient ischaemic attack, amaurosis fugax, cardiovascular death (according to Swedish National Registers)
Number of participants suffering post-operative cardiovascular events (by 2027) | Follow up assessment year 2027 (recording of events occurring since 2025)
  Post-operative myocardial infarction, stroke, transient ischaemic attack, amaurosis fugax, cardiovascular death (according to Swedish National Registers)
Number of participants suffering post-operative cardiovascular events (by 2029) | Follow up assessment year 2029 (recording of events occurring since 2027)
  Post-operative myocardial infarction, stroke, transient ischaemic attack, amaurosis fugax, cardiovascular death (according to Swedish National Registers)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Goncalves, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Skåne University Hospital (SUS), Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
No sharing allowed due to General Data Protection Regulation (GDPR) legislation as sensitive personal data is included.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT05821894/Prot_SAP_001.pdf